CLINICAL TRIAL: NCT04254068
Title: Preventing Feeding and Eating Disorders in Children of Parents With Eating Disorders: A Randomized Controlled Trial
Brief Title: Parent-Based Prevention (PBP) for Parents With Eating Disorders
Acronym: PBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, James Dale Lock, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29032
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Eating Disorders; Eating Behavior
Keywords: Secondary prevention; Parent-based prevention
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomized case series trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent based prevention (Experimental): Parent-Based Prevention (PBP; Sadeh-Sharvit & Lock, 2018) is a manualized preventive intervention, focused on increasing parental awareness and competence to facilitate healthy eating habits, body image, and self-regulation in children whose parent has an eating disorder history. PBP is comprised of three phases that focus on unique goals. The strategies in each session include psycho-education, behavioral experiment planning, and skill practicing to augment parents' insight into how the context of the parental cognitions and behaviors may impact child outcomes, with the goal of creating a longstanding effect.
  Interventions: Behavioral: Parent-based prevention
- Usual care (No Intervention): Families randomized to usual care will be permitted to utilize any medical, psychological, or nutritional services they desire for the waitlist period of 16 weeks.

INTERVENTIONS:
Behavioral: Parent-based prevention — Parent-based prevention is a 12 session program for parents with eating disorders and their partners. Most sessions occur on a weekly basis, most of the sessions involve both partners.
  Other Names: PBP
  Arms: Parent based prevention

SUMMARY:
Parents with eating disorders exhibit greater concerns and dilemmas about developing healthy habits in their children. Studies indicate that the offspring of parents with eating disorders have more developmental and interpersonal difficulties. Consequently, these parents should receive personalized care to enhance their parental capacity and support them in their decision making process. The Parent-Based Prevention of Eating Disorders (PBP) is a promising intervention that may help improve feeding and eating practices and children outcomes, by engaging both parents in a short-term program. This study aims to empirically evaluate the feasibility and acceptability of PBP over a wait-list control group (i.e., treatment-as-usual) in a Randomized Case Series Trial.

DETAILED DESCRIPTION:
A parental history of an eating disorder is linked with greater risk of eating and socio-emotional problems in the offspring, and more stressful parent-child interactions. Further, parenting concerns often exacerbate existing eating disorder symptoms in parents. Parent-Based Prevention (PBP-B) is a focused intervention aimed to support parents with eating disorders and their partners in developing healthy eating and lifestyle behaviors in their children. The program also focuses on reducing mealtime conflict and improving couple communication. This study tests the feasibility, acceptability and preliminary outcomes of the Parent-Based Prevention (PBP) program for these parents and their partners. Parents with any lifetime eating disorder diagnosis who have at least one child 1-5 years old will be randomized to receive PBP immediately or following a 16-week waitlist period. This study will investigate whether PBP is feasible, acceptable, and associated with improvement in short-term outcomes that predict long term risks of eating and weight disorders (e.g., parental cognition associated with feeding practices and child eating behaviors and socio-emotional symptoms). The study will collect important case series data that will inform the design of larger, adequately powered studies to test ways to reduce the likelihood of eating and weight difficulties in the offspring of parents with eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* A biological parent of a child between 1-5 years of age.
* A lifetime diagnosis of an eating disorder.

Exclusion Criteria:

* Current medical condition necessitating more intensive care to manage symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting parents with a lifetime diagnosis of an eating disorder: Number of eligible participants that agree to participate in the study | Up to 48 months
  Number of eligible participants that agree to participate in the study
Acceptability of the intervention: Client Satisfaction Questionnaire score | Week 12
  Mean Client Satisfaction Questionnaire score at end of treatment. Scores range on a Likert-like scale of 1-5, with higher scores indicative of greater satisfaction.

SECONDARY OUTCOMES:
Parental feeding practices | Baseline and Week 12
  Change scores of the Child Feeding Questionnaire from baseline to end of treatment. Scores range on a Likert-like scale of 1-5, with higher scores indicative of the parent endorsing more frequent behaviors on the dimension measured.
Child eating behaviors | Baseline and Week 12
  Change scores of the Children's Eating Behavior Questionnaire from baseline to end of treatment. Scores range on a Likert-like scale of 1-4, with higher scores indicative of greater endorsement of the behavior measured.

CONTACTS AND LOCATIONS:
Overall Officials: Shiri Sadeh-Sharvit, PhD, Principal Investigator — s
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No